CLINICAL TRIAL: NCT03032718
Title: Effects of Individually Tailored Whole-body Vibration Training on the Symptoms of Chemotherapy-induced Peripheral Neuropathy: a Randomized-controlled Trial
Brief Title: Whole-body Vibration Training to Reduce the Symptoms of Chemotherapy-induced Peripheral Neuropathy
Acronym: VANISH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Basel (Other)
Collaborators: German Sport University, Cologne (Other); University Hospital of Cologne (Other); University of Freiburg (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Oliver Faude, Deputy Head Exercise and Movement Science, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-01527
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding against study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will receive a defined exercise program twice a week in addition to their usual treatment. Training sessions start immediately after randomization and will be supervised by trained sport students. They will take place twice a week, for twelve weeks in specific training rooms designed to meet the needs of oncological patients in the respective centers. The vibration exercises will take place on a side-alternating vibration platform (GalileoTM, Pforzheim, Germany) ®) according to the previously determined optimal (highest neuromuscular response) setting for each individual. Each session will last for about 15 to 30 minutes, leaving sufficient time for regeneration. Training will consist of four vibration exercises, chosen from a standardized pool of exercises with increasing difficulty in order to allow for individual, optimal progression. All sessions will be documented by the supervisor.
  Interventions: Behavioral: Whole-body vibration training
- Control (No Intervention): Patients in the control group will receive treatment as usual and will be given the opportunity to participate in the intervention after completion of the study.

INTERVENTIONS:
Behavioral: Whole-body vibration training — Whole-body vibration exercise
  Arms: Intervention

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a highly prevalent and clinically meaningful side effect of cancer treatment. It is induced by neurotoxic chemotherapeutic agents, causing severe sensory and/or motor deficits such as pain, altered sensation, reduced or absent reflexes, muscle weakness, reduced balance control, insecure gait, and higher risk of falling. It is associated with significant disability and poor recovery, not only reducing patients' autonomy and quality of life but also limiting medical cancer therapy, which subsequently may affect the clinical outcome and compromise survival. To date, CIPN cannot be prevented and approved and effective treatment options are lacking.

Promising results regarding CIPN have recently been achieved with exercise. Own preliminary work revealed that patients profit from sensorimotor training (SMT), experiencing significant relief from CIPN induced symptoms. In a pilot study we therefore also evaluated whole body vibration training, a further neuromuscular stimulating exercise intervention. Results suggest that whole body vibration (WBV) is not only feasible and safe for neuropathic cancer patients but can attenuate motor and sensory deficits.

We therefore propose a two-armed, multicenter, randomized controlled trial (RCT with a follow-up period), including 44 patients with neurologically confirmed CIPN, in order to evaluate the effects of WBV on the relevant symptoms of CIPN. Primary endpoint is the patient reported reduction of CIPN-related symptoms (FACT-GOG-Ntx). Secondary endpoints will include compound muscle action potentials, distal motor latency, conduction velocity, and F-waves from the tibial and peroneal nerve as well as antidromic sensory nerve conduction studies of the sural nerve, feasibility, non-invasive electromyographic (EMG) activity of mm. tibialis anterior, soleus, gastrocnemius medialis, rectus femoris, vastus medialis and biceps femoris, peripheral deep sensitivity, proprioception, balance control as well as pain, quality of life and the level of physical activity. Patients will be assessed before and after a 12 week intervention and again after 12 weeks of follow-up. Interim tests will be performed 6 weeks into the intervention as well as every 3 weeks during the follow-up.

We hypothesize that individually tailored whole body vibration training will reduce relevant symptoms of CIPN. Our results could contribute to improve supportive care in oncology, thereby enhancing patients' quality of life and coincidentally enabling the optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* oncological patients with neurologically confirmed CIPN
* age: 18-80 years
* performance status of 0-2 according to the toxicity and response criteria of the Eastern Cooperative Oncology Group
* patients underwent neurotoxic chemotherapy with one of the following agents: Taxanes (docetaxel with a cumulative dose of ≥ 225mg/m2 or paclitaxel with a cumulative dose of ≥ 525mg/m2), Vinca-alkaloids (vincristine with a cumulative dose of ≥ 4.2mg/m2 or vinblastine with a cumulative dose of 24mg/m2), Platinum-derivatives (Oxaliplatin with a cumulative dose of ≥ 510mg/m2, Cisplatinum with a cumulative dose of ≥ 200mg/m2)

Exclusion Criteria:

* pre-existing neuropathy of other cause (e.g. diabetes)
* given contraindications for WBV (instable osteolysis, osteosynthesis, acute thrombosis, foot ulcers and a fracture of a lower extremity in the last two years)
* a myocardial infarction, angina pectoris or heart disease (NYHA III-IV) within the past six months
* a mental condition or lack of the German language that prevents the understanding of the written informed consent
* metastases of the central nervous system and epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG-Ntx questionnaire [Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity] | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  It will be used to document and assess the severity of the subjective peripheral neuropathy (PNP) symptoms. This questionnaire has been validated and is widely applied in clinical practise. It contains eleven items which allow an assessment of the extent of PNP symptoms - from "not at all" to "very much".

SECONDARY OUTCOMES:
Compound muscle action potentials (CMAP) | Baseline
  obtained from the tibial and peroneal nerve
Distal motor latency | Baseline
  obtained from the tibial and peroneal nerve
Nerve conduction velocity | Baseline
  obtained from the tibial and peroneal nerve
Sensory nerve action potentials (SNAPs) | Baseline
  recorded from the lateral malleolus with surface electrodes
Peripheral deep sensitivity | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  evaluated with a Rydel-Seiffer tuning fork (128Hz) on a scale from 0 to 8; due to age related neural deconditioning, values ≤4 are pathological for patients ≥ 60years old, while for patients under 60 years old, ≤5 is regarded as pathological
Reflex action | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  The Achilles tendon reflex as well as the patellar tendon reflex is assessed with a reflex hammer and graded on a 3 point scale (1=agile, 2=weak, 3=missing).
Sense of position | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  This test examines whether patients can recognize a change of position in their first toe, with their eyes closed.
Perception of touch | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  The examiner symmetrically strokes the outsides of the patients' legs and feet in order to detect reduced or altered sensation due to demyelination or axonal degeneration.
Muscular strength | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  The strength of the leg muscles is assessed by requesting the patient to actively move their legs against the resistance of the examiner's arm. The examiner then grades the strength on a six point scale (0=no activity, 1=visual contraction without motor effect, 2=movement under elimination of gravity, 3=movement under gravity, 4=movement against slight resistance 5=normal force).
EMG recordings | 1 week (first 2 training sessions)
  Normalized (to static standing without vibration condition) integrated EMG activity of mm. tibialis anterior, soleus, gastrocnemius (medial head), mm. rectus femoris, vastus medialis, biceps femoris. EMG recordings will be performed using bipolar Ag/AgCl surface electrodes placed over the mm. soleus, gastrocnemius medialis, tibialis anterior, rectus femoris, vastus medialis and biceps femoris of the right leg. A reference electrode will be placed on the patella. To keep interelectrode resistance below 2 kOhm, the skin areas for the electrodes will have to be shaved, degreased and slightly abraded. The EMG signals will then be transmitted to the amplifier (band-pass filter 10 Hz-1 kHz, 1,0009 amplified) via shielded cables and recorded with 4 kHz.
CIPN-related pain | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  Visual analogue scale (VAS) in order to assess neuropathic pain as well as the dysesthesias
Postural control | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
  Center of pressure during upright static and dynamic stance
Quality of life - questionnaire | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up
Physical activity questionnaire | Change over the course of the study, from baseline to post 12-week intervention to post 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Streckmann, PhD, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Streckmann F, Hess V, Bloch W, Decard BF, Ritzmann R, Lehmann HC, Balke M, Koliamitra C, Oschwald V, Elter T, Zahner L, Donath L, Roth R, Faude O. Individually tailored whole-body vibration training to reduce symptoms of chemotherapy-induced peripheral neuropathy: study protocol of a randomised controlled trial-VANISH. BMJ Open. 2019 Apr 24;9(4):e024467. doi: 10.1136/bmjopen-2018-024467. PMID 31023750